CLINICAL TRIAL: NCT04717128
Title: Evaluation of Health Professional Learners' Competence in Newborn Positioning and Attachment Following a Standardized Patient-led Lactation Skills Workshop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LiquidGoldConcept (Industry)
Collaborators: University of Michigan (Other); Michigan State University (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 21-002
Record Dates: First submitted 2021-01-05; First posted 2021-01-20 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Breastfeeding; Patient Simulation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Participants will be cluster randomized to complete the standardized-patient led breastfeeding skills workshop with one of the baby dolls.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Standardized patients leading the workshop will know which baby doll they are using in the workshop. Participants will not know whether or not they are receiving "treatment" and investigators and data analysts will be blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baby doll with user remote controlled jaw (Experimental): In this arm, standardized patients will use the Newborn Oral Assessment and Latch Simulator (NORALSim) to demonstrate and teach newborn positioning and attachment in the breastfeeding skills workshop.
  Interventions: Other: Breastfeeding Skills Workshop
- Baby doll with hand controlled jaw (Active Comparator): In this arm, standardized patients will use a cloth baby doll with a puppet-style mouth to demonstrate and teach newborn positioning and attachment in the breastfeeding skills workshop.
  Interventions: Other: Breastfeeding Skills Workshop

INTERVENTIONS:
Other: Breastfeeding Skills Workshop — Participants will complete the standardized patient-led breastfeeding skills workshop where they will learn breast massage techniques to alleviate plugged ducts and engorgement, hand expression of breast milk, effective breast pump use, and newborn positioning and attachment.

SUMMARY:
Evaluating newborn positioning and attachment is a key skill for maternal-child healthcare providers. Trainees have limited opportunities to practice this skill in their clinical rotations due to a lack of access to lactating patients. Thus, positioning and attachment training is traditionally conducted through passive modalities, primarily videos.

Investigators aim to evaluate the impact of an interactive breastfeeding skills workshop using a baby doll on health professional learners' ability to identify effective and ineffective positioning and attachment at the breast.

DETAILED DESCRIPTION:
Faculty at the University of Michigan School of Public Health (UM-SPH), Johns Hopkins School of Nursing (JHUSON), and Michigan State University (MSU) are collaborating with LiquidGoldConcept (LGC), a company focusing on simulation-based training in maternal-child care, to evaluate the impact of high-fidelity simulation on health professional learner outcomes. For the Phase I SBIR, LGC is developing a high-fidelity newborn simulator for healthcare professional education in clinical lactation.

Evaluating newborn positioning and attachment is a key skill for maternal-child healthcare providers. Trainees have limited opportunities to practice this skill in their clinical rotations due to a lack of access to lactating patients. Thus, positioning and attachment training is traditionally conducted through passive modalities, primarily videos.

Investigators aim to evaluate the impact of an interactive breastfeeding skills workshop using a baby doll on health professional learners' ability to identify effective and ineffective positioning and attachment at the breast.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in a health professional training program (e.g. medical student, nursing student, physician resident)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
(Pre-Intervention) Competence in Evaluating Newborn Positioning and Attachment | Day 1 (Pre-Intervention)
  Participants will complete a pre-intervention knowledge check on newborn positioning and attachment prior to and immediately following the Breastfeeding Skills Workshop. The knowledge check will consist of 5 true-false questions. For each question, the participant will watch a 3-second clip of positioning and attachment and respond to the question "True or False, I would recommend adjustments to this dyad's positioning and attachment." For each true/false question, participants will respond to a multiple-choice question with 4 options on why they would or would not make adjustments to the dyad.
(Post-Intervention) Competence in Evaluating Newborn Positioning and Attachment | Day 1 (Post-Intervention)
  Participants will complete a post-intervention knowledge check on newborn positioning and attachment prior to and immediately following the Breastfeeding Skills Workshop. The knowledge check will consist of 5 true-false questions. For each question, the participant will watch a 3-second clip of positioning and attachment and respond to the question "True or False, I would recommend adjustments to this dyad's positioning and attachment." For each true/false question, participants will respond to a multiple-choice question with 4 options on why they would or would not make adjustments to the dyad.

SECONDARY OUTCOMES:
Performance of Clinical Lactation Skills related to positioning and attachment in a Video-based Simulation (Telesimulation) | 1-12 weeks
  The Standardized Patient in that telesimulation will rate their performance of clinical and communication skills using a 10-item Formative Assessment Rubric (FAR). The FAR includes four "I know" statements rating clinical skills specific to the case scenario (e.g. I know why my nipples have been hurting when I breastfeed my baby).
Performance of Clinical Lactation Skills related to positioning and attachment in a Video-based Simulation (Telesimulation) | 1-12 weeks
  An independent rater will watch audio-video recordings of the telesimulation and grade learner's completion of technical skills relevant to positioning and attachment according to a 14-point checklist (Point values: 0=did not complete, 1=did complete)
Satisfaction with the Breastfeeding Skills Workshop | 1-12 weeks
  Participants will complete a 6-item satisfaction survey immediately following completion of the second telesimulation with the following items. Participants will rate their agreement on a 6-point Likert scale (1=strongly disagree, 6=strongly agree)
  1. The skills workshop helped me prepare for the positioning and attachment telesimulation.
  2. The multiple-choice questions helped me prepare for the positioning and attachment telesimulation.
  3. What was expected of me as a health professional during the telesimulation was appropriate for my level of training.
  4. The amount of time allotted for the telesimulation was adequate.
  5. The standardized patient in the telesimulation was a realistic breastfeeding mother.
  6. The newborn simulator distracted from the realism of the telesimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- LiquidGoldConcept, Ypsilanti, Michigan, United States

IPD SHARING:
Plan to Share IPD: No